CLINICAL TRIAL: NCT04642729
Title: Fresh Corneal Lenticule Implantation in Macular Corneal Distrophy With Relex-Smile Surgery
Brief Title: Fresh Corneal Lenticule Implantation in Macular Corneal Distrophy With Relex Smile Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EyeHP
Record Dates: First submitted 2020-11-20; First posted 2020-11-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Macular Corneal Dystrophy
MeSH Terms: conditions — Corneal Dystrophies, Hereditary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReLex Smile surgery (Other): The myopic lenticule after Relex Smile surgery is put into BBS solution for 10 min. Under topical anesthesia, Using VisuMax Femtosecond Laser.
  Interventions: Procedure: Fresh Corneal Lenticule Implantation using Relex-Smile Surgery
- fresh corneal lenticule implantation (Other): Using VisuMax Femtosecond Laser we make intrastromal pocket incision 2-3 mm in periphery of cornea (Because the macular dystrophy is in the center more progressive) and 150 µm deep to put fresh corneal lenticule. After one month using VisuMax we create a flap using autologous serum with purpose to remove more dead keratocytes and adding live keratocytes with aim to regenerate the metabolism of cornea.
  Interventions: Procedure: Fresh Corneal Lenticule Implantation using Relex-Smile Surgery

INTERVENTIONS:
Procedure: Fresh Corneal Lenticule Implantation using Relex-Smile Surgery — Knowing that the most important element is damage of stroma we used all preoperative procedures atlas, optic tomography and especially electron microscope. Approximately we planned how much microns we remove and insert, for example we remove 80 µm and we insert fresh corneal lenticule 90 µm with the purpose to remove more dead keratocytes which increase biomechanical instability of corneal metabolism (abnormal increase collagenase activity, decrease proteinase inhibitors, excessive premature keratocyte apoptosis, increase cytokine binding). Fresh Corneal Lenticule and autologous serum contains live stem cells that produce keratocytes, collagen fibers, extracellular matrix which contribute to the regeneration of the cornea, and all this results at increasing of corneal transparency and visual acuity in patients with corneal macular dystrophy.
  Other Names: Relex smile surgery

SUMMARY:
The aim of the study is to examine the effect of fresh corneal lenticule implantation as allogenic graft taken from myopic patients to implanted in patients with macular corneal dystrophy using Visumax Femtosecond Laser Smile module surgery.

DETAILED DESCRIPTION:
Macular Corneal Dystrophy is a severe form of stromal corneal dystrophy characterized by bilateral cloudy regions within hazy stroma and eventually severe visual impairment.

Most cases of MCD are caused by mutations in the CHST6 gene encoding a protein involved in the production of keratan sulfate, which plays a role in the maintenance of corneal transparency.

According to biomechanical instability of corneal metabolism (abnormal increase collagenase activity, decrease proteinase inhibitors, excessive premature keratocyte apoptosis, increase cytokine binding) at corneal dystrophies. Fresh Corneal Lenticule and autologous serum contains live stem cells that produce keratocytes, collagen fibers, extracellular matrix which contribute to the regeneration of the cornea, and all this results at increasing of corneal transparency and visual acuity in patients with corneal macular dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* indications for penetrating keratoplasty
* low transparec of corneae
* low visual acuity

Exclusion Criteria:

* active anterior segment pathology
* previous corneal or anterior segment surgery
* any infection

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Increase of corneal transparency | 12 months
  Implanting fresh corneal lenticule we add more live stem cells and keratocytes to stabilize biomechanical stability of cornea. Also making flap and putting autologous serum after one month of implanting fresh corneal lenticule we removed more dead keratocytes from macula dystrophia and added more live keratocytes which contributed to the regeneration of the cornea.

SECONDARY OUTCOMES:
Increase of visual acuity | 12 months
  After implanting fresh corneal lenticule according to clarity of cornea visual acuity increased for 2-3 m and also softening symptoms of corneal dystrophy ex. dry eyes, sensitivity to light, pain in the eye, corneal erosion etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo